CLINICAL TRIAL: NCT03431675
Title: Cluster-randomized Trial to Evaluate the Impact of Ciprofloxacin Prophylaxis as a Response to a Meningococcal Meningitis Epidemic
Brief Title: Ciprofloxacin for the Prevention of Meningococcal Meningitis 2018
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: No epidemic of Men C in 2019
Sponsor: Epicentre (Other)
Collaborators: Medecins Sans Frontieres, Netherlands (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Cipro chemoprophylaxis 2018
Record Dates: First submitted 2018-02-06; First posted 2018-02-13 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Meningitis, Meningococcal
MeSH Terms: conditions — Meningitis, Meningococcal | interventions — Ciprofloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard care (No Intervention): No chemoprevention for contacts of cases of meningitis (current standard of care) with a health promotion visit by a study nurse after the first notification of cases during the epidemic
- Household prophylaxis arm (Active Comparator): Chemoprophylaxis with a single dose of oral ciprofloxacin for household members of reported cases of meningitis. For participants age >12 years: 500 mg tablet; age 5-12 years: 250 mg tablet; age 1-4 years: 125 mg tablet; age 3-11 months: 100 mg (2 ml oral suspension); age <3 months: 75 mg (1.5 ml oral suspension)
  Interventions: Drug: Ciprofloxacin
- Community prophylaxis arm (Active Comparator): Chemoprophylaxis with ciprofloxacin in the setting of a village-wide distribution after the notification of the first case of meningitis in a village. For participants age >12 years: 500 mg tablet; age 5-12 years: 250 mg tablet; age 1-4 years: 125 mg tablet; age 3-11 months: 100 mg (2 ml oral suspension); age <3 months: 75 mg (1.5 ml oral suspension)
  Interventions: Drug: Ciprofloxacin

INTERVENTIONS:
Drug: Ciprofloxacin — Single-dose oral ciprofloxacin
  Other Names: Cipro
  Arms: Community prophylaxis arm; Household prophylaxis arm

SUMMARY:
The trial is an interventional, cluster-randomized trial to assess the impact of oral ciprofloxacin for household and community contacts of meningitis cases on the incidence of meningitis during an epidemic.

The trial contains a nested sub-study ("resistance study") to assess the effect of a single dose of ciprofloxacin on the prevalence of fluoroquinolone-resistant enterobacteriaceae in the study area.

DETAILED DESCRIPTION:
The study is designed as a cluster-randomized trial in the setting of a meningitis epidemic to assess the impact of chemoprophylaxis with single-dose ciprofloxacin on the incidence of meningitis in the study area.

The study will be implemented in a health district in Niger where a meningitis outbreak is occurring, and where Médecins Sans Frontières is providing assistance to the Ministry of Health in its outbreak response. In order to launch the study protocol, at least two Health Areas (HA) of a Health District (HD) will have met the weekly epidemic threshold of 10 cases per 100 000 per week, or of 5 cases per week if the population of the HA is less than 30 000 people, following the most recent WHO recommendations for meningitis surveillance.

All villages in the HAs which have crossed the epidemic threshold and are included in the study area will be randomized to receive standard care, household-level prophylaxis or community-wide prophylaxis.

Once a HA has been included in the study, a case-based surveillance system will be put in place, or reinforced if one is currently in place in the study area. Suspected cases of meningitis that present to health posts will be referred to the nearest health center. In each health center, the diagnosis and treatment of meningitis will follow national protocols.

In the standard care arm, after the first case has been notified from a village, a study nurse will visit the village with a local community member. The study nurse will lead an informational session for members of the community regarding the signs and symptoms of meningitis, and the urgency of presenting to the nearest health center as soon as possible if any of those signs or symptoms arrive. In the household-level prophylaxis arm, each time a case is reported from a village that has been randomized to this arm, a study nurse will visit the household of the notified case within 24 hours. The study nurse will offer ciprofloxacin to all persons currently living in the same household compound and present at the time of the visit. In the community-level prophylaxis arm, after the first case is reported from a village that has been randomized to this arm, a member of study staff will visit the village within 24 hours. During this visit, arrangements will be made for a community-wide distribution of ciprofloxacin, preferably within 72 hours of the initial case presentation at the health center / district hospital. A series of informational meetings will be organized before the distribution.

If the epidemic is in an urban setting, neighborhoods will be randomized to one of the three arms in a 1:1:1 ratio. If the epidemic is in a rural area, villages will be randomized to either standard care or village-wide prophylaxis in a 1:1 ratio.

A nested substudy to assess the effects of ciprofloxacin prophylaxis on the prevalence of ciprofloxacin-resistant enterobacteriaceae will be carried out among 400 persons (200 in the standard care arm and 200 in the community-wide prophylaxis arm). Participants will provide a series of 3 stool samples for culture, speciation, and antibiotic resistance testing.

ELIGIBILITY:
Inclusion Criteria:

* Resident in a village included in the study area

Exclusion Criteria:

* Patients currently exhibiting symptoms of meningitis (to be immediately referred for further care)
* Persons with a known allergy to fluoroquinolone antibiotics.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-03-01 (Estimated); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Meningitis attack rate | From enrollment of a village through study completion, an average of 2 months
  The primary outcome aims to evaluate the impact of a chemoprevention strategy as a public health intervention during a meningitis outbreak, which is best evaluated by looking at the overall attack rates in the study area.

SECONDARY OUTCOMES:
Proportion of participants with ciprofloxacin-resistant enterobacteriaceae in their stools | Prior to ciprofloxacin dosing (day 0) and at 7 and 28 days post-ciprofloxacin dosing
  A substudy is proposed to compare rates of acquisition of ciprofloxacin resistance among participants in the standard care arm and participants in the village prophylaxis arm. 20 participants in 10 villages in each of the two arms will be asked to provide stool samples on days 0, 7 and 28
Proportion of patients who received ciprofloxacin who develop meningitis | From enrollment of a village through study completion, an average of 2 months
  This secondary outcome aims to evaluate the impact of a chemoprevention strategy as a public health intervention during a meningitis outbreak, which is best evaluated by looking at the overall attack rates in the study area.
Meningitis attack rate by sex | From enrollment of a village through study completion, an average of 2 months
  This secondary outcome aims to evaluate the impact of a chemoprevention strategy as a public health intervention during a meningitis outbreak, which is best evaluated by looking at the overall attack rates in the study area.
Meningitis attack rate by age | From enrollment of a village through study completion, an average of 2 months
  This secondary outcome aims to evaluate the impact of a chemoprevention strategy as a public health intervention during a meningitis outbreak, which is best evaluated by looking at the overall attack rates in the study area.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca F GRAIS, PhD, Study Director — Epicentre
Locations (1):
- Madarounfa Health District, Madarounfa, Maradi Region, Niger

IPD SHARING:
Plan to Share IPD: Yes
A de-identified data set can be made available after the signature of an appropriate data sharing agreement.